CLINICAL TRIAL: NCT05196477
Title: Multicentre Non-interventional Retrospective Cohort Study of the Outcomes of Olokizumab Therapy in Hospitalized Patients With SARS-CoV-2 (COVID-19) Infection
Brief Title: Study of the Outcomes of Olokizumab Therapy in Hospitalized Patients With SARS-CoV-2 (COVID-19) Infection
Acronym: ROCOVI
Status: Completed | Type: Observational
Sponsor: R-Pharm (Industry)
Collaborators: Almedis LLC (Unknown); Data Management 365 (Industry); ScienceFiles LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: CL04041090
Record Dates: First submitted 2022-01-18; First posted 2022-01-19 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; 2019-nCoV; Severe acute respiratory syndrome coronavirus 2; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — olokizumab; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Olokizumab treatment group: Subjects with the infection caused by SARS-CoV-2 who received olokizumab injection in addition to the standard therapy.
  Interventions: Drug: Olokizumab; Drug: Standard therapy
- Standard treatment group: Subjects with the infection caused by SARS-CoV-2 who received the standard therapy without monoclonal antibodies (mAbs).
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Olokizumab — The details of taking olokizumab, including its route of administration, dose and frequency of taking the drug as part of routine clinical practice, will be registered in the electronic case report forms (eCRFs).
  Groups: Olokizumab treatment group
Drug: Standard therapy — Standard treatment (excluding administration of olokizumab, other interleukin (IL) (interleukin-1 and interleukin-17) inhibitors and Janus-kinase inhibitors.

SUMMARY:
The study purpose was to assess the outcomes of therapy with olokizumab within complex therapy of Coronavirus disease 2019 (COVID-19) in hospitalised patients in real clinical practice setting. The study investigated patients' characteristics, disease progression, and efficacy and safety of olokizumab therapy.

DETAILED DESCRIPTION:
This was a multicentre retrospective cohort study of patients admitted to hospitals in various Russian Federation cities with positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) nucleic acid (RNA) laboratory test for the treatment of severe acute respiratory syndrome. The study used information from primary medical documentation of COVID-19 patients who had underwent diagnostic and therapeutic procedures in accordance with the hospital clinical practice. Clinical and laboratory data was collected and analysed to assess olokizumab safety, investigate other treatments, course and outcomes of the disease.

No additional tests or medical procedures were made as part of this study. If any data collected under the protocol was not available or not collected, they deemed lacking.

Based on the results of preliminary assessment of the number of records from the patients meeting inclusion / exclusion criteria in the clinical sites planning to participate in the project it was planned to include no more than 3000 patients in the study, of which about 1500 would be in the main group (received olokizumab therapy), and 1500 would be in the comparison group. It was planned to conduct an analysis in the general population (including taking into account its balancing using statistical methods, in case of significant differences in the initial characteristics of patients in groups), as well as in a subpopulation selected from pairs formed taking into account the comparability of patients by individual characteristics. In total, it was planned to form at least 200 pairs (or more, if the included population is highly comparable). Participation of several clinics in Russian Federation cities (not more than 10 cites) was expected to assure sufficient population for the study.

Data collection period for each hospitalised patient was equivalent to in-hospital period for the treatment of SARS-CoV-2 infection. Data collection by patients was made during hospital stay, including the day of discharge (treatment outcome or lethal outcome). The primary study variables were defined during 21-day observation period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SARS-CoV-2 (using virus ribonucleic acid polymerase chain reaction (RNA PCR) test).
* Hospital admission for COVID-19 therapy.
* Infiltrative lung changes based on imaging findings (chest X-ray, chest computed tomography (CT)).
* Indications for Preemptive anti-inflammatory therapy (PAT), including two or more signs below:

  * reduced oxygen saturation of the blood SpO2 ≤ 97 %
  * C-reactive protein (CRP) > 15 mg/L
  * body temperature > 37.5 °C for at least 3 days
  * white blood cell count < 4.0 x 10^9/L
  * absolute lymphocyte count < 2.0 x 10^9/L.
* Olokizumab therapy - for the test group.
* Source medical documents contain the information required for the study (lacking or incomplete data on some serum chemistry values are allowed: D-dimer, ferritin, IL-6, procalcitonin).

Exclusion Criteria:

* Inadequate information on patient's characteristics and therapy.
* Lack of documented confirmation of SARS-CoV-2 infection.
* Initiation of mechanical ventilation (MV) from the first day of admission in the control group or before olokizumab administration in the test group.
* Administration of systemic corticosteroids, IL-6, other immunosuppressants or immunoglobulins before hospital admission.
* Lack of indications to PAT
* Administration of olokizumab, other interleukin (IL) (interleukin-1 and interleukin-17) inhibitors and Janus-kinase inhibitors - for comparator group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study enrolls males and females aged ≥ 18 years with infection caused by SARS-CoV-2 who received in-hospital therapy. The study population includes all the patients admitted to hospital since June 2020, meeting inclusion / exclusion criteria with their data collected and analysed.
Sampling Method: Probability Sample
Enrollment: 3087 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who died during hospital admission due to any reason | up to 21 days
  The percentage of patients who died during hospital admission due to any reason in each therapy group

SECONDARY OUTCOMES:
The percentage of patients who required mechanical ventilation or transfer to intensive care unit (ICU), or who died during hospital admission due to COVID-19 | up to day 21
  The percentage of patients who required mechanical ventilation or transfer to ICU, or who died after olokizumab therapy during hospital admission due to COVID-19.
The percentage of patients who required transfer to ICU | up to day 21
  The percentage of patients who required transfer to ICU in each therapy group
The percentage of patients who required transfer to a new type of oxygen support and to an invasive mechanical ventilation (MV) | up to day 21
  The transfer to a new type of oxygen support means the transfer to a more severe type of oxygen support (the appointment of low-current oxygen to patients who were initially without oxygen support; transfer from low-flow oxygen therapy to high-flow, non-invasive or invasive ventilation; from high-flow oxygen therapy to non-invasive or invasive ventilation; from non-invasive to invasive ventilation).
Overall hospitalisation period | from admission to discharge from hospital, up to 21 days
  Overall hospitalisation period duration in each therapy group (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (6):
- Russia (6):
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University" under the Ministry of Health of the Russian Federation, Kazan', Tatarstan Republic
  - Federal State Budgetary Educational Institution of Higher Education Bashkir State Medical University of the Ministry for Healthcare of the Russian Federation, Ufa, The Republic of Bashkortostan
  - State Budgetary Healthcare Institution "Regional Hospital № 3", Chelyabinsk
  - State Budgetary Healthcare Institution "City Clinical Hospital named after F.I. Inozemtsev of Moscow Healthcare Department", Moscow
  - St. Petersburg State Budgetary Healthcare Institution "City Hospital No. 40 of the Kurortny District", Saint Petersburg
  - State Budgetary Institution of Healthcare of Tver region "Regional clinical hospital", Tver'